CLINICAL TRIAL: NCT00717808
Title: A Phase 1, Blinded, Randomised, Crossover Pilot Study to Investigate the Safety, Tolerability and Pharmacokinetics of Tranilast in Patients With Rheumatoid Arthritis on Methotrexate
Brief Title: Effects of Tranilast on Pharmacokinetics of Methotrexate (MTX) in Patients With Rheumatoid Arthritis (RA)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to unforeseen circumstances this study will not now start.
Sponsor: Imperial College London (Other)
Collaborators: Nuon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112007; 2007-005357-39 (EudraCT Number); REC Ref:08/H0707/2 (Other: Ethics Committee); R&D ref: TAYP2010 (Other: University Identifier)
Record Dates: First submitted 2008-07-14; First posted 2008-07-18 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2011-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Tranilast; Rheumatoid Arthritis; Pharmacokinetics; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tranilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): During the study the patient will either receive tranilast (300mg twice a day) or a placebo drug for a period of seven days. The patient will then have a seven day break followed by another period of seven days in which the patient will receive the other medication.
  Interventions: Drug: Tranilast
- 2 (Placebo Comparator): The patient will receive the placebo twice a day for 7 days whilst taking their weekly methotrexate dose
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Tranilast — Tranilast (300mg twice a day) for a period of seven days whilst taking their weekly prescribed dose of methotrexate. Followed by a 7 day washout period before starting arm 2
  Other Names: Rizaben (Tranilast); 3',4'-dimethoxycinnamonyl anthranilic acid
  Arms: 1
Drug: Placebo comparator — The patient will receive the placebo capsule twice a day whilst receiving their weekly dose of methotrexate
  Other Names: Lactose Monohydrate
  Arms: 2

SUMMARY:
The treatment of rheumatoid arthritis has improved considerably in recent years with the understanding that better outcomes can be achieved by optimising the dosage schedule of conventional drugs that suppress the inflammatory response in joints. Furthermore, the development of protein based drugs that are given parenterally (i.e. by subcutaneous injection or intravenous infusion), known as biologics, have given rise to even better clinical results. However, despite this over 60% of patients with rheumatoid arthritis can still be expected to have an unacceptably high degree of disease activity and the prohibitively high cost of biologic therapy has resulted in rationing following NICE review. Therefore there is a need for more effective and less costly treatment.

The proposed study is designed to test potential drug interactions between one such candidate oral treatment, tranilast, and the gold standard therapy for rheumatoid arthritis, methotrexate, which is given as a once weekly oral, intramuscular or intradermal regimen. The drug to be tested, tranilast, an analogue of a naturally occurring molecule that regulates inflammatory responses, is currently used in the treatment of allergic inflammation and has recently been shown to be effective in an animal model of multiple sclerosis. Tranilast is an analogue of a naturally tryptophan metabolite. Laboratory studies of cell biology indicate that this molecule inhibits a number of key inflammatory pathways and the function of white blood cells that play a critical role in the inflammatory features of rheumatoid arthritis. The aim of this study is to assess whether tranilast may be useful for the treatment of RA. In an animal model of rheumatoid arthritis, initial assessment showed that prophylactic administration of tranilast interfered with the development of disease. Therapeutically, in an animal model of arthritis, tranilast was very effective, and reduced all aspects of the disease, including joint swelling, clinical score, and histological damage in a dose-dependent fashion, and reduced pain. This degree of benefit compares well with therapeutics that have been highly successful in humans, such as anti-TNF therapy. Furthermore studies at the Kennedy Institute of Rheumatology Division, Imperial College suggest that tranilast has a greater analgesic effect than the potent steroid dexamethasone at effective anti-inflammatory doses

DETAILED DESCRIPTION:
THEORETICAL FRAMEWORK:The treatment outcomes in rheumatoid arthritis have dramatically improved with the recognition that the inflammatory component of disease needs to be suppressed optimally at every stage in its evolution. However, all existing conventional oral therapies are associated with limited efficacy and loss of effectiveness over time. Furthermore all of these therapies are associated with significant toxicity and tolerability problems. Another approach to treatment involves the use of biologic (protein based), parenterally administered therapies directed against important inflammatory molecules or cells involved in disease pathology. Despite the notable success of anti-TNF therapy, which is one of these biologics,approximately one third of patients do not respond adequately and the costs of drug production are very high.

This causes rationing in all healthcare economies. There is therefore a need for new, safe, well tolerated and effective drugs that are cost effective. Tranilast (a tryptophan metabolite) is already licenced in Japan for the treatment for allergy. Basic science studies including those undertaken at The Kennedy Institute indicate that this drug suppresses the activity of a number of key inflammatory mediators as well as the activation of lymphocytes (white blood cells) responsible for the perpetuation of inflammation and associated tissue destruction in rheumatoid. Therefore, there was a rationale to test the effectiveness of tranilast in vivo for the treatment of arthritis. In an animal model of arthritis, tranilast effectively reduces joint swelling and read outs of pain. Since tranilast is well tolerated and safe in the licenced treatment indication in man, it is timely to test its effectiveness in rheumatoid arthritis. The majority of patients with this condition are treated with methotrexate often in combination with other anti-rheumatoid drugs. The current study is a prelude to a larger randomised controlled study investigating the efficacy of tranilast in rheumatoid arthritis.

PURPOSE:This study will evaluate the pharmacokinetics, safety and tolerability of an oral medication, tranilast, in patients with rheumatoid arthritis who are on another disease modifying medication, methotrexate.

DESIGN:The study is a randomised crossover pilot study with an optional higher dose open label phase.

METHOD:During the study the patient will either receive tranilast (300mg twice a day) or a placebo drug for a period of seven days. The patient will then have a seven day break followed by another period of seven days in which the patient will receive the other medication. They will attend the clinic on at least 6 occasions(screening, day 2,3 8 and 9 then on 5 occasions in session 2 plus a follow up session. During the study blood samples will be taken to assess safety and serum concentrations of the study drug and interactions with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and non-pregnant, non-lactating women between 18 and 75 years of age. Sexually active females must be of either non-childbearing potential or willing to comply with the contraceptive requirements.
* Body weight greater >40 kg and <120 kg with a body mass index (BMI) between 19-31 kg/m2
* Clinical history of rheumatoid arthritis as defined by ACR criteria and currently on a stable dosing regimen of methotrexate 7.5 to 25 mg once weekly, as their only DMARD (no changes in dosing regimen for 4 weeks prior to screening).
* Negative urine pregnancy test (for all women except those with documented proof of hysterectomy or bilateral oophorectomy)
* Subjects who are able and willing to give written consent

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening history, physical exam, clinical laboratory evaluations or ECG, with the exception of values related to rheumatoid arthritis.
* Estimated Glomerular Filtration rate <60mL/min.
* Significant hepatic insufficiency as defined by total bilirubin greater than 25.7umol/L or transaminase(ALT, AST) elevations greater than 2 times the upper limit of the clinical laboratory range. Also any patient with documented cirrhosis or a history consistent with a diagnosis of cirrhosis or hepatitis.
* Patients not on a stable DMARD and/or NSAID drug regimen, or expecting to remain on a stable drug regimen, as defined by starting a new drug or changing dosage within 14 days prior to administration of study medication.
* Patients taking any drugs known to be substrates of CYP2C9 or taking digoxin, or cerivastatin within 14 days prior to Session 1, or taking any drugs known to inhibit or induce CYP2C9.
* Known or suspected hypersensitivity to tranilast or to structurally similar compounds.
* History of recurrent urinary tract infections or kidney stones.
* History of an acute illness within 2 weeks prior to the first dose of study medication.
* History of alcohol abuse within 2 years preceding the first dose of study medication.
* History of gout or hyperuricaemia.
* History of drug abuse within 2 years preceding the first dose of study medication.
* Use of an investigational drug within 30 days preceding the first dose of study medication.
* Donation of blood in excess of 500 mL within 56 days prior to the first dose of study medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Plasma pharmacokinetics of tranilast and methotrexate following multiple doses of tranilast in patients with Rheumatoid Arthritis. | Predosing on day 8 and throughout day 8 and 24 hours later on day 9 for both sessions 1 and 2

SECONDARY OUTCOMES:
Safety and tolerability of tranilast in combination with methotrexate will also be assessed | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Taylor, PhD, Principal Investigator — Imperial College London

REFERENCES:
- [Background] Platten M, Ho PP, Youssef S, Fontoura P, Garren H, Hur EM, Gupta R, Lee LY, Kidd BA, Robinson WH, Sobel RA, Selley ML, Steinman L. Treatment of autoimmune neuroinflammation with a synthetic tryptophan metabolite. Science. 2005 Nov 4;310(5749):850-5. doi: 10.1126/science.1117634. PMID 16272121
- [Background] Inglis JJ, Criado G, Andrews M, Feldmann M, Williams RO, Selley ML. The anti-allergic drug, N-(3',4'-dimethoxycinnamonyl) anthranilic acid, exhibits potent anti-inflammatory and analgesic properties in arthritis. Rheumatology (Oxford). 2007 Sep;46(9):1428-32. doi: 10.1093/rheumatology/kem160. Epub 2007 Jul 21. PMID 17644821